CLINICAL TRIAL: NCT03168542
Title: Clinical Evaluation of Fitting Investigational Contact Lenses Phase 2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johnson & Johnson Vision Care, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR-5955
Record Dates: First submitted 2017-05-22; First posted 2017-05-30 (Actual); Results first posted 2018-10-19 (Actual); Last update posted 2018-10-19 (Actual); Status verified 2018-09

CONDITIONS: Visual Acuity

STUDY DESIGN:
Intervention Model Description: While this study utilizes two contact lenses, the purpose was to evaluate the JJVC fitting guide. This was a non-randomized study in which eye care practitioners used the JJVC fitting guide to fit subjects with a study contact lens. Subjects may fit either in a bilateral or a contralateral fashion.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Toric Multifocal Contact Lens (Experimental): JJVC Investigational Toric Multifocal Contact Lens for Presbyopia
  Interventions: Device: JJVC Fitting Guides
- Multifocal Contact Lens (Experimental): 1-Day Acuvue® Moist Brand Multifocal Contact Lens
  Interventions: Device: JJVC Fitting Guides

INTERVENTIONS:
Device: JJVC Fitting Guides — Subjects who are habitual soft spherical or toric contact lens wearers, at least 40 years of age and no more than 70 years of age, will be fitted, according to the fitting guide, with either the Multifocal Contact Lens or an Investigational Toric Multifocal Contact Lens if refractive cylinder power of the eye is between -1.00 to -1.50. The Intervention is approximately 30-90 minutes during a 1 day visit.

SUMMARY:
This study is a single arm, non-randomized, open label, bilateral, non- dispensing clinical trial with only one visit. The Eye Care Providers will be provided with a fitting guide and will determine the initial study lens selection. Each subject will wear either the investigational contact lenses or marketed contact lenses for approximately 30-90 minutes. This study aims to evaluate the ECPs impression of the fitting guide for a novel multifocal lens and also their success in fitting the lenses.

ELIGIBILITY:
Inclusion Criteria:

1. The subject must read, understand, and sign the STATEMENT OF INFORMED CONSENT and receive a fully executed copy of the form.
2. The subject must appear able and willing to adhere to the instructions set forth in this clinical protocol.
3. Healthy adult males or females that are at least 40 years of age and no more than 70 years of age.
4. The subject must either be wearing a presbyopic contact lens correction (e.g., reading spectacles over contact lenses, multifocal or monovision contact lenses, etc.) or if not respond positively to at least one symptom on the "Presbyopic Symptoms Questionnaire".
5. The subject is a current soft spherical or toric contact lens wearer (defined as a minimum of 6 hours of wear per day at least two days of the week for a minimum of 1 month prior to the study).
6. The subject's distance spherical equivalent or spherical component (if the eye has - 1.00 to -1.50 D of refractive cylinder) of their refraction must be in the range -1.25 D to -3.75 D or +1.25 D to +3.75 D in each eye.
7. The subject's refractive cylinder cannot be greater than -1.50D in either eye.
8. The subject's refractive cylinder axis must be 90°±30° or 180°±30° in each eye.
9. The subject's ADD power must be in the range of +0.75 D to +2.50 D in each eye.
10. The subject must have best corrected visual acuity of 20/20-3 or better in each eye.
11. The subject must have a wearable pair of spectacles if required for their distance vision.

Exclusion Criteria:

1. Ocular or systemic allergies or disease, or use of medication which might interfere with contact lens wear.
2. Pregnancy or lactation.
3. Currently diagnosed with diabetes.
4. Infectious diseases (e.g. hepatitis, tuberculosis) or an immune-suppressive disease (e.g. HIV).
5. Clinically significant (Grade 3 or 4) corneal edema, corneal vascularization, corneal staining, tarsal abnormalities or bulbar injection, or any other corneal or ocular abnormalities which would contraindicate contact lens wear.
6. Entropion, ectropion, extrusions, chalazia, recurrent styes, dry eye, glaucoma, history of recurrent corneal erosions.
7. Any previous, or planned, ocular or intraocular surgery (e.g., radial keratotomy, PRK, LASIK, lid procedures, cataract surgery, retinal surgery, etc.).
8. A history of amblyopia, strabismus or binocular vision abnormality.
9. Any ocular infection or inflammation.
10. Any ocular abnormality that may interfere with contact lens wear.
11. Use of any ocular medication, with the exception of rewetting drops.
12. History of herpetic keratitis.
13. Participation in any contact lens or lens care product clinical trial within 30 days prior to study enrollment.
14. Employee of clinical site (e.g., Investigator, Coordinator, Technician)

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2017-05-01 (Actual); Primary Completion 2017-05-04 (Actual); Study Completion 2017-05-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Vistakon Research Clinic, Jacksonville, Florida, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 23 subjects were enrolled into this study. Of the enrolled subjects 21 were dispensed a study lens and 2 subjects failed to meet the eligibility criteria. Of the dispensed subjects all 21 completed the study.
Pre-assignment Details: This was a non-randomized study. The JJVC fitting guide, subjects responses and eye car practitioner options dictated which study lens the subject was to be fit with. Lens type and lens sequence are not experimental design factors. The first lens pair (Right/Left) on eye was the same lens pair (Right/Left) the subject ended with.
Groups:
- Toric Multifocal/Toric Multifocal: Subjects that wore the Toric Multifocal contact lens in both eyes (Right/Left) for the entire duration of the study.
- Toric Multifocal/ Multifocal: Subjects that wore the Toric Multifocal contact lens in their right eye and the Sphere Multifocal contact lens in their left eye for the entire duration of the study.
- Multifocal/Toric Multifocal: Subjects that wore the Sphere Multifocal contact lens in their right eye and the Toric Multifocal contact lens in their left eye for the entire duration of the study.
Period: Overall Study
Arm/Group | Toric Multifocal/Toric Multifocal | Toric Multifocal/ Multifocal | Multifocal/Toric Multifocal
Started | 7 | 5 | 9
Completed | 7 | 5 | 9
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Dispensed Subjects: All subjects dispensed at least one study lens.
Arm/Group | Dispensed Subjects
Number analyzed (Participants) | 21
Age, Continuous [Mean (Standard Deviation); unit: Years] | 57.0 (6.05)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18
  Male | 3
Race/Ethnicity, Customized [Number; unit: Participants]
  Black or African American | 4
  White | 17
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 21

OUTCOME MEASURES:

1. Primary Outcome: Number of Fitting Modifications to Optimize Vision
Description: The ECP followed the fitting guide to assess the vision provided by the study lenses and determined if a lens change was needed. The ECP modified the lenses based upon the subject's responses in accordance with the Fitting Guide. Two modifications were allowed. The number of modifications required by the ECP to optimize vision was recorded.
Time Frame: 15 Minutes Post Lens Fitting
Population: All subjects that completed the study without a major protocol deviation.
Measure: Mean (Standard Deviation); unit: Lens
Units Other Than Participants: Eyes
Groups:
- JJVC Fitting Guides: ECPs used JJCV Fitting guides to fit subjects with the Toric Multifocal contact lens in both eyes and the Sphere Multifocal contact lens in both eyes.
Arm/Group | JJVC Fitting Guides
Number analyzed (Participants) | 21
Number analyzed (Eyes) | 42
Lens | 0.21 (0.47)
Statistical Analysis 1: Comparison: JJVC Fitting Guides; Test type: Superiority — Superiority was concluded if the lower 95% of the confidence limit of the proportion of subjects who require no more than one modification was greater than 50%; Agresti-Coull confidence interval; Agresti-Coull method was used to estimate the confidence interval of the binomial proportions; Proportion = 0.952, 95% CI 2-sided [0.756 to 1.000]

2. Secondary Outcome: Subject's Responses to Individual Item 1
Description: Subjects responses to individual item "Considering Your Experience With The Study Contact Lenses, Which Statement Best Describes Your Overall Satisfaction Of These Contact Lenses?". This item had a response set of extremely satisfied, very satisfied, moderately satisfied, slightly satisfied and not at all satisfied. The percentage of subject's in each response category was reported.
Time Frame: 15 Minutes Post Lens Insertion
Population: All subjects that completed the study without a major protocol deviation.
Measure: Number; unit: Percentage of participants
Arm/Group | JJVC Fitting Guides
Number analyzed (Participants) | 21
Percentage of participants
  Extremely satisfied | 23.8
  Very satisfied | 66.7
  Moderately satisfied | 4.8
  Slightly satisfied | 4.8
  Not at all satisfied | 0

3. Secondary Outcome: Subject's Responses to Individual Item 2
Description: Subjects responses to individual item "Based On Your Experience Today, How Likely Are You To Purchase This Contact Lens?". This item had a response set of extremely likely, very likely, somewhat likely, slightly likely and not at all likely. The percentage of subject's in each response category was reported.
Time Frame: 15 Minutes Post Lens Insertion
Population: All subjects that completed the study without a major protocol deviation
Measure: Number; unit: Percentage of participants
Arm/Group | JJVC Fitting Guides
Number analyzed (Participants) | 21
Percentage of participants
  Extremely likely | 33.3
  Very likely | 52.4
  Somewhat likely | 9.5
  Slightly likely | 0
  Not at all likely | 4.8

4. Secondary Outcome: Subject's Responses to Individual Item 3
Description: Subjects responses to individual item "Please Think About Your Experience Today With The Study Contact Lenses. Please Indicate How You Satisfied You Are With The Overall Contact Lens Fitting Process?". This item had a response set of very satisfied, satisfied, unsure, dissatisfied and very dissatisfied. The percentage of subject's in each response category was reported
Time Frame: 15 Minutes Post Lens Insertion
Population: All subjects that completed the study without a major protocol deviation.
Measure: Number; unit: Percentage of participants
Arm/Group | JJVC Fitting Guides
Number analyzed (Participants) | 21
Percentage of participants
  Very Satisfied | 66.7
  Satisfied | 28.6
  Unsure | 4.8
  Dissatisfied | 0
  Very Dissatisfied | 0

5. Secondary Outcome: Subject's Responses to Individual Item 4
Description: Subjects responses to individual item "Where Would You Expect To Go Looking For Information About This Contact Lens? Please Select All That Apply.". The percentage of subject's in each response category was reported.
Time Frame: 15 Minutes Post Lens Insertion
Population: All subjects that completed the study without a major protocol deviation.
Measure: Number; unit: Percentage of participants
Arm/Group | JJVC Fitting Guides
Number analyzed (Participants) | 21
Percentage of participants
  On a website for particular brand of contacts | 71.4
  On a general healthcare website such as WebMD | 9.5
  In a Magazine | 19.1
  In a Newspaper | 9.5
  On a search engine (ex: Google) | 42.9
  On a Blog | 4.8
  On Social Media Networks | 19.1
  On YouTube | 9.5
  In an Online Forum | 4.8
  On your Vision Care Insurance Website | 23.8
  Talking with friends family or colleagues | 47.6
  Talking with an eye doctor | 81.0
  Online, but not through an advertisement | 23.8
  Other | 4.8

6. Secondary Outcome: Subject's Responses to Individual Item 5
Description: Subjects responses to individual item "If You Were To Purchase The Study Contact Lenses, With What Frequency Would You Expect To Wear Them?". This item had a response set of All of the time, Usually, Frequently, Sometimes, Rarely and never. The percentage of subject's in each response category was reported.
Time Frame: 15 Minutes Post Lens Insertion
Population: All subjects that completed the study without a major protocol deviation.
Measure: Number; unit: Percentage of participants
Arm/Group | JJVC Fitting Guides
Number analyzed (Participants) | 21
Percentage of participants
  All of the time | 85.7
  Usually | 9.5
  Frequently | 4.8
  Sometimes | 0
  Rarely | 0
  Never | 0

7. Secondary Outcome: Subject's Responses to Individual Item 6
Description: Subjects responses to individual item "What Are Your Current Vision Correction Solutions?". The percentage of subject's in each response category was reported.
Time Frame: 15 Minutes Post Lens Insertion
Population: All subjects that completed the study without a major protocol deviation.
Measure: Number; unit: Percentage of participants
Arm/Group | JJVC Fitting Guides
Number analyzed (Participants) | 21
Percentage of participants
  Toric Contact Lenses | 23.8
  Multifocal Contact Lenses | 52.4
  Monovision | 23.8
  Readers | 28.6
  Progressive Lenses | 19.1
  Other | 4.8

8. Secondary Outcome: Subject's Responses to Individual Item 7
Description: Subjects responses to individual item "How did the new lens you tried as a part of this clinical study Compare To Your Current Vision Correction Solutions?". This item had a response set of Much better, somewhat better, about the same, somewhat worse and much worse. The percentage of subject's in each response category was reported.
Time Frame: 15 Minutes Post Lens Insertion
Population: All subjects that completed the study without a major protocol deviation.
Measure: Number; unit: Percentage of participants
Arm/Group | JJVC Fitting Guides
Number analyzed (Participants) | 21
Percentage of participants
  Much better | 42.9
  Somewhat better | 28.6
  About the same | 19.1
  Somewhat worse | 9.5
  Much worse | 0

9. Secondary Outcome: Subject's Responses to Individual Item 8
Description: Subjects responses to individual item "Considering your experience with the study contact lens, how excited are you about this lens being available to purchase?". This item had a response set of Very Excited, Excited, Unsure, Unexcited and Very Unexcited. The percentage of subject's in each response category was reported.
Time Frame: 15 Minutes Post Lens Insertion
Population: All subjects that completed the study without a major protocol deviation.
Measure: Number; unit: Percentage of participants
Arm/Group | JJVC Fitting Guides
Number analyzed (Participants) | 21
Percentage of participants
  Very Excited | 42.9
  Excited | 38.1
  Unsure | 14.3
  Unexcited | 4.8
  Very Unexcited | 0

10. Secondary Outcome: Subject's Responses to Individual Item 9
Description: Subjects responses to individual item "How would you rate your overall visual performance with the study contact lens?". This item had a response set of Excellent, Very Good, Good, Fair and Poor. The percentage of subject's in each response category was reported.
Time Frame: 15 Minutes Post Lens Insertion
Population: All subjects that completed the study without a major protocol deviation.
Measure: Number; unit: Percentage of participants
Arm/Group | JJVC Fitting Guides
Number analyzed (Participants) | 21
Percentage of participants
  Excellent | 33.3
  Very Good | 57.1
  Good | 4.8
  Fair | 4.8
  Poor | 0

11. Secondary Outcome: Subject's Responses to Individual Item 10
Description: Subjects responses to individual item "Considering Your Experience With The Study Contact Lenses, Which Statement Best Describes Your Overall Opinion Of These Contact Lenses?". This item had a response set of Excellent, Very Good, Good, Fair and Poor. The percentage of subject's in each response category was reported.
Time Frame: 15 Minutes Post Lens Insertion
Population: All subjects that completed the study without a major protocol deviation.
Measure: Number; unit: Percentage of participants
Arm/Group | JJVC Fitting Guides
Number analyzed (Participants) | 21
Percentage of participants
  Excellent | 38.1
  Very Good | 52.4
  Good | 4.8
  Fair | 4.8
  Poor | 0

ADVERSE EVENTS:
Time Frame: Throughout the entire duration of the study. Approximately 1 day per subject.
Groups:
- Toric Multifocal: Subjects that wore the Toric Multifocal contact lens at any point during this study.
- Multifocal: Subjects that wore the Sphere Multifocal contact lens at any point during this study.
Arm/Group | Toric Multifocal | Multifocal
All-Cause Mortality (participants affected / at risk) | 0/21 | 0/14
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/14
Other Adverse Events (participants affected / at risk) | 0/21 | 0/14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-04-17): https://cdn.clinicaltrials.gov/large-docs/42/NCT03168542/Prot_SAP_000.pdf